CLINICAL TRIAL: NCT06684028
Title: PET Image Exploration of Novel Tracer [68Ga]-FAPI-JNU Imaging Studies in Patients with Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2024013
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Solid Malignancies
Keywords: FAP; FAPI; PET; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI-JNU (Experimental): 68Ga-FAPI-JNU is administered through a superficial vein on the back of the hand. A PET/CT scan was performed approximately 1 hour after injection
  Interventions: Drug: 68Ga-FAPI-JNU

INTERVENTIONS:
Drug: 68Ga-FAPI-JNU — Patients will receive the novel tracer 68Ga-FAPI-JNU dose of approximately 2-5 mCi per person

SUMMARY:
To investigate the biological distribution of a new tracer 68Ga-FAPI-JNU in the primary, metastatic and normal tissues of patients with malignant tumors, and to evaluate the biological distribution of 68GA-FAPI-JNU with standardized uptake values.

DETAILED DESCRIPTION:
PET/CT imaging was performed about 1 hour after the patient was injected with the novel tracer 68Ga-FAPI-JNU. SUVmax and SUVmean values of the area of interest were mapped by two diagnostic physicians with more than 5 years of experience after the imaging was completed.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects sign the informed consent voluntarily and can complete the test according to the protocol requirements;
2. Age 18-85 years old, male or female;
3. Clinically diagnosed as malignant tumor, diagnostic criteria refer to biopsy or other imaging such as CT and MRI;
4. ECOG score is 0-3 points;

Exclusion Criteria:

1. Patients with a history or allergic constitution to any component of the developer, including alcohol;
2. pregnant or lactating women;
3. Patients with mental illness or related history;
4. Patients who cannot or cannot undergo a PET/CT scan;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the distribution of 68Ga-FAPI-JNU in tumors, metastases and normal tissues | 4 hour
  CT and PET scans were performed on the patients injected with 68Ga-FAPI-JNU. After image reconstruction and PET/CT image fusion, the biological distribution of 68Ga-FAPI-JNU in the primary tumor, metastatic tumor and various tissues and organs of the patients was evaluated by radioactive uptake value (standardized uptake value, SUV)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiated Hospital of Jiangnan University, Wuxi, Jiangsu, China